CLINICAL TRIAL: NCT04518839
Title: The Comparison of Cognitive Function, Symptoms of Depression and Anxiety, and Quality of Life in Patients After Hip Fracture Surgery Under General or Regional Anesthesia
Brief Title: The Comparison of Cognition, Depression and Anxiety, and Quality of Life After Hip Fracture Surgery Under General or Regional Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Tea Fabijanić, MD, MD, University of Zagreb
Other Study IDs: 643-03/20-07/33,380-130/134-20
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Cognitive Dysfunction; Hip Fractures; Depression, Anxiety; Quality of Life
Keywords: hip fracture surgery; regional anaesthesia; general anaesthesia; postoperative cognitive dysfunction; depression; anxiety; quality of life
MeSH Terms: conditions — Postoperative Cognitive Complications; Hip Fractures; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with regional anaesthesia
- Group with general anaesthesia

SUMMARY:
Postoperative cognitive dysfunction is a relatively common in elderly patients after hip surgery, but exact mechanism of its onset is still unclear as well as contributing factors. There is also increased incidence of depression and anxiety. Both affect the recovery after surgery, slow it down and reduce the quality of life. Patients will be divided into two groups, operated under regional anaesthesia and operated under general anaesthesia, and monitored after surgery. Patients will be tested before and after surgery to evaluate postoperative cognitive deficits, depression and anxiety scale and health-related quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients intended for surgical treatment of hip fractures ≥ 60 years
* Patients who are category ASA I to ASA III will be included in research
* Sufficient cognitive ability
* Only those patients who have agreed to be participants in the research and have signed the consent for participation and informed consent.

Exclusion Criteria:

* Patients who refused to participate in the survey and who did not sign informed consent
* Patients with ASA IV or more
* Patients under 60 years
* Severe psychiatric disorders involving the use of psychopharmaceuticals back three months
* All patients who have other fractures in addition to hip fractures
* Polytrauma
* All patients scheduled for more than one surgical intervention during the procedure, or within the next 8 weeks
* Patients who have been diagnosed with dementia, and / or are receiving anti-dementia drugs

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical treatment of hip fractures in Clinical Hospital Center Zagreb.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
change in cognition | preoperatively/postoperative follow up 2 months
  MoCA scale (Montreal Cognitive Assessment), F-A-S test
change in anxiety and depression | preoperatively/postoperative follow up 2 months
  The HAD Scale (The Hospital Anxiety and Depression Scale)
change in quality of life | preoperatively/postoperative follow up 2 months
  EQ-5D-5L Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tea Fabijanić, MD, Principal Investigator — University of Zagreb